CLINICAL TRIAL: NCT04426565
Title: The 9-month Follow-up Study for the Patients of Illicit Substance Use Disorder After Receiving the Different Psychosocial Intervention
Brief Title: The Follow-up Study for the Patients of Illicit Substance Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Kai-Suan Psychiatric Hospital (Other Government)
Collaborators: Kaohsiung Medical University (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSPH-2019-23
Record Dates: First submitted 2020-05-19; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Substance Use Disorders; Illicit Drug Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The motivational enhancement interview, the individual psychotherapy, the group psychotherapy, the family therapy will be provided by our team members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- the motivational enhancement interview (Other): The motivational enhancement interview is a counseling approach developed in part by clinical psychologists William R. Miller and Stephen Rollnick. It is a directive, client-centered counseling style for eliciting behavior change by helping clients to explore and resolve ambivalence.
  Interventions: Behavioral: the individual psychotherapy; Behavioral: the group psychotherapy; Behavioral: the family therapy
- the individual psychotherapy (Other): The individual psychotherapy is the use of psychological methods, particularly when based on regular personal interaction with adults, to help a person change behavior and overcome problems in desired ways. Psychotherapy aims to improve an individual's well-being and mental health, to resolve or mitigate troublesome behaviors, beliefs, compulsions, thoughts, or emotions, and to improve relationships and social skills.
  Interventions: Behavioral: motivational enhancement interview; Behavioral: the group psychotherapy; Behavioral: the family therapy
- the group psychotherapy (Other): The group psychotherapy is a form of psychotherapy in which one or more therapists treat a small group of clients together as a group. The term can legitimately refer to any form of psychotherapy when delivered in a group format, including Art therapy, cognitive behavioural therapy or interpersonal therapy, but it is usually applied to psychodynamic group therapy where the group context and group process is explicitly utilised as a mechanism of change by developing, exploring and examining interpersonal relationships within the group.
  Interventions: Behavioral: motivational enhancement interview; Behavioral: the individual psychotherapy; Behavioral: the family therapy
- the family therapy (Other): The family therapy is is a branch of psychotherapy that works with families and couples in intimate relationships to nurture change and development. It tends to view change in terms of the systems of interaction between family members.
  Interventions: Behavioral: motivational enhancement interview; Behavioral: the individual psychotherapy; Behavioral: the group psychotherapy

INTERVENTIONS:
Behavioral: motivational enhancement interview — Motivational interviewing is supported by over 200 randomized controlled trials across a range of target populations and behaviors including substance abuse, health-promotion behaviors, medical adherence, and mental health issues.
  Arms: the family therapy; the group psychotherapy; the individual psychotherapy
Behavioral: the individual psychotherapy — It has been demonstrated to be an effective treatment for depression and has been modified to treat other psychiatric disorders such as substance use disorders and eating disorders. It is incumbent upon the therapist in the treatment to quickly establish a therapeutic alliance with positive countertransference of warmth, empathy, affective attunement and positive regard for encouraging a positive transferential relationship, from which the patient is able to seek help from the therapist despite resistance.
  Arms: the family therapy; the group psychotherapy; the motivational enhancement interview
Behavioral: the group psychotherapy — Group psychotherapy is a key component of milieu therapy in a therapeutic community. The total environment or milieu is regarded as the medium of therapy, all interactions and activities regarded as potentially therapeutic and are subject to exploration and interpretation, and are explored in daily or weekly community meetings. A form of group therapy has been reported to be effective in psychotic adolescents and recovering addicts.
  Arms: the family therapy; the individual psychotherapy; the motivational enhancement interview
Behavioral: the family therapy — According to a 2004 French government study conducted by French Institute of Health and Medical Research, family and couples therapy was the second most effective therapy after Cognitive behavioral therapy. The study used meta-analysis of over a hundred secondary studies to find some level of effectiveness that was either "proven" or "presumed" to exist. Of the treatments studied, family therapy was presumed or proven effective at treating schizophrenia, bipolar disorder, anorexia and substance dependence.
  Arms: the group psychotherapy; the individual psychotherapy; the motivational enhancement interview

SUMMARY:
The patients will be diagnosed according to DSM-5, the severity of individual substance use disorder will be assessed, and the plan of treatment will be provided. The treatment will be determined by the diagnosis and severity of addiction, the mood or psychiatric comorbidities, the hyperactivity or attention deficit, alcohol addiction, and etc. The motivational enhancement interview, the individual psychotherapy, the group psychotherapy, the family therapy will be provided by our team members. In order to evaluate the efficacy of the different therapy, we will evaluate the psychological and social status of the patients and follow up every 3 months. The efficacy of different treatment will be evaluated according to our study instruments.

DETAILED DESCRIPTION:
The patients will be diagnosed according to DSM-5, the severity of individual addiction will be assessed, and the plan of treatment will be provided. The treatment will be determined by the diagnosis and severity of addiction, the mood or psychiatric comorbidities, the hyperactivity or attention deficit, alcohol addiction, and etc. The motivational enhancement interview, the individual psychotherapy, the group psychotherapy, the family therapy will be provided by our team members. In order to evaluate the efficacy of the different therapy, we will evaluate the psychological and social status of the patients and follow up every 3 months.

The patients will be received the basic physiological assessment, the chest X-ray, electrocardiogram, liver and renal function, hematology test, urine screening for addictive substances, screening for blood infectious diseases (including hepatitis B, C and HIV infection) will be included.

Besides, the Drug Abuse Screen Test (DAST), the Severity of Dependence Scale (SDS), the Reliability of Readiness to Change Questionnaire, the Opiate Treatment Index (OTI), drug Avoidance Self-Efficacy Scale (DASES), the Family APGAR score, The brief version of the World Health Organization Quality of Life instrument (WHOQOL-BREF Taiwan version), Chinese health questionnaire (CHQ), parental bonding instrument (PBI), Toronto Alexithymia Scale (TAS), Brief Symptom Rating Scale (BSRS-5), Chinese version of Adult ADHD Self-Report Scale (ASRS-V1. 1), Becker Depression Scale (BDI) and Becker Anxiety Scale (BAI) will be evaluated every 3 months after receiving our treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients with illicit substance use disorder diagnosed by DSM-5

Exclusion Criteria:

The age of the patient is below 20 years old or above 65 years old, the patients cannot cooperate with the tools of investigation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
The severity of substance use used by the Severity of Dependence Scale | 9 months
  The value is from 0 to 15, and higher scores mean a worse outcome.
The World Health Organization Quality of Life instrument (WHOQOL-BREF Taiwan version) | 9 months
  The instrument has four dimension and higher scores mean a better outcome.
Becker Depression Scale | 9 months
  The value is from 0 to 63, and higher scores mean a worse outcome.
Becker Anxiety Scale | 9 months
  The value is from 0 to 63, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Huang-Chih Chou, Ph.D., Principal Investigator — Kaohsiung Municipal Psychiatric Hospital
Locations (1):
- Kaohsiung Municipal Kai-Syuan Psychiatric Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No